CLINICAL TRIAL: NCT04049487
Title: Targeted Exercise in a Group Setting Compared to General Group Fitness Class: Impact on Diastasis Recti in Postpartum Women
Brief Title: Impact of Exercise on Diastasis Rectus Abdominus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Y Stone, Manager, Clinical Rehabilitative Services, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016673
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Diastasis Recti and Weakness of the Linea Alba
Keywords: postpartum; diastasis recti; diastasis rectus
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be matched and randomly assigned to two groups: a general exercise group and a diastasis specific group. Each group will participate in a 4 week long exercise program.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be matched and sorted by a non clinical research staff member. The participant will not know which group they are in, nor will the outcomes assessor. The people who are leading the 2 exercise groups will know which the groups are, but will take care not to mention to participants which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generalized Exercise (Active Comparator): General wellness/exercise program designed to replicate a generic wellness program that one would find in a gym setting. Will be led by an exercise instructor.
  Interventions: Other: Exercise
- Diastasis Specific Exercise (Experimental): Diastasis specific exercise program incorporating multiple muscle groups and based on research findings of exercises that are shown to be effective for reducing size and impact of diastasis rectus.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups will participate in group exercise as previously described

SUMMARY:
The aim with this research project is to evaluate the success of diastasis recti closure after a 4-week group exercise class that includes: strengthening of each abdominal muscle group, hip strengthening and stabilization, and pelvic floor activation and cueing during exercises. Success will be evaluated by measuring width and depth of linea alba laxity before and after completion of the 4 sessions as well as other outcome measures such as lumbopelvic pain, pain with intercourse, and incontinence. Intervention will be compared to a control group that participates in an exercise program geared toward general health and wellness.

DETAILED DESCRIPTION:
Diastasis recti, is a condition where the linea alba becomes stretched, sometimes lax, and creates distance between the rectus abdominis muscle bellies. It occurs most often during and after pregnancy, abdominal weight gain, and sometimes due to straining while performing heavy lifting. If the linea alba becomes thin enough to tear, the person may experience a hernia. Inter-rectus distance >25mm (~2 finger widths) at one or more locations is considered to be clinically significant for diastasis recti. Pathological diastasis recti is an inter rectus distance widening more than 10mm (~1 finger width) above the umbilicus, 27mm (~2.5 finger widths) at the umbilicus, and 9mm (~1 finger width) below the umbilicus. Normal width of the linea alba in nulliparous women should be less than 15mm at the xiphoid process, 22 mm at 3cm above the umbilicus, and 16mm at 2 cm below umbilicus.

The prevalence of diastasis recti is significant in the postpartum population. Clinically significant diastasis recti is currently thought to be best assessed at 2cm above the umbilicus and 5cm above the umbilicus between 25-41 weeks of pregnancy, and at 6 months postpartum. At 6 months postpartum, the average values for diastasis recti using these measurements were 23mm average at 2cm above the umbilicus (~2.5 finger widths), and 18mm average at 5cm above the umbilicus (~2 finger widths). The measures below the umbilicus were clinically insignificant at 6 months postpartum.

Thed abdominal drawing-in maneuver (transverse abdominis activation) and curl up (rectus abdominis activation) are both exercise maneuvers that have been traditionally taught for diastasis resolution. It was found that curl ups alone narrow the inter-rectus distance but don't achieve tension through the linea alba. Transverse abdominis activation alone tensions the linea alba but doesn't achieve narrowing of the inter-rectus distance. Combined transverse abdominis activation and curl up achieves both narrowing and tension through the linea alba.

The positive correlation between diastasis recti and lumbopelvic pain, incontinence, and pelvic organ prolapse has been shown in recent studies as well. 52% of urogynecological patients had a diastasis recti in one study, and that 66% of those women had a support-related pelvic floor dysfunction (i.e. stress urinary incontinence (UI), fecal incontinence (FI), and/or pelvic organ prolapse (POP)). 45% of women in pregnancy have pelvic girdle pain (PGP), and 25% in the early postpartum period still have PGP. 5-7% of women continue to experience PGP at 12 wks postpartum. 45% of women have urinary incontinence at 7 years postpartum; 27% of those who were initially incontinent in the early postpartum period regained continence, but 31% who were initially continent became incontinent by 7 years postpartum, thus highlighting the need for early intervention of postpartum rehab.

In recent years, research on diastasis recti has become more prevalent. However, the research on diastasis recti recovery and physical therapy treatment programs is limited. Most of the studies thus far have looked at transverse abdominis activation, curl ups, and planks. Effects of strengthening abdominal obliques, hips, pelvic floor, and heavier strengthening of the rectus abdominis done at the same time have not yet been included in these studies.

The aim with this research project is to evaluate the success of diastasis recti closure after a 4-week group exercise class that includes: strengthening of each abdominal muscle group, hip strengthening and stabilization, and pelvic floor activation and cueing during exercises. Success will be evaluated by measuring width and depth of linea alba laxity before and after completion of the 4 sessions as well as other outcome measures such as lumbopelvic pain, pain with intercourse, and incontinence. Intervention will be compared to a control group that participates in an exercise program geared toward general health and wellness.

The goal is to evaluate whether a program incorporating hip, core, and pelvic floor strengthening specifically designed to address the weaknesses common in individuals with diastasis recti is superior to a generalized wellness program in addressing lumbopelvic pain, incontinence, and other pelvic health conditions. If so, this will lay the foundation for a protocol to guide the clinician on safe, yet effective, methods of core strengthening so women are able to transition back into community fitness classes safely and without fear of worsening their diastasis recti.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Has had a vaginal or cesarean delivery between 12 weeks and 2 years ago
* Has a diastasis measured at least 2 cm wide

Exclusion Criteria:

* Cardiovascular problems precluding exercise
* Exercise-induced asthma
* History of stroke
* History of abdominal surgery other than a cesarean section
* Current pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Diastasis width comparison | At enrollment (prior to intervention), within 1 week following end of intervention
  Measured by the same outcomes assessor, reported in centimeters
Diastasis depth comparison | At enrollment (prior to intervention), within 1 week following end of intervention
  Measured by the same outcomes assessor, reported in centimeters

SECONDARY OUTCOMES:
Back pain comparison | At enrollment (prior to intervention), within 1 week following end of intervention
  Measured using the Numeric Pain Rating scale. This scale measures pain on a spectrum from 0 (no pain) to 10 (worst pain you can imagine) and is validated for use in comparison within an individual.
Incontinence comparison | At enrollment (prior to intervention), within 1 week following end of intervention
  Measured by presence or absence, frequency of leaking, need for pads
Dyspareunia comparison | At enrollment (prior to intervention), within 1 week following end of intervention
  Using the Marinoff Dyspareunia Scale Score. This scale measures level of dyspareunia (pain with sex) on a spectrum from 0 (no limitations to sex) to 3 (unable to participate in penetrative intercourse due to pain).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y Stone, DPT, Principal Investigator — University of Missouri Health Care
Locations (1):
- MU Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Only the person who is doing data input will have access to IPD.